CLINICAL TRIAL: NCT05583383
Title: A Phase II Clinical Study of the New Adjuvant Treatment of HER-2 Positive Resectable Locally Advanced Adenocarcinoma of Stomach and Gastroesophageal Junction With Camrelizumab+SOX Control Camrelizumab+SOX+ Trastuzumab
Brief Title: A Study of the Advanced Adenocarcinoma of Stomach and Gastroesophageal Junction With Camrelizumab+SOX Control Camrelizumab+SOX+ Trastuzumab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, LiuYing, Chief physician, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-GC-002
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): camrelizumab was administered intravenously at a fixed dose of 200 mg, on the first day, once every 3 weeks, with a cycle of 3 weeks. Infusion for 30 min each time (no less than 20 min and no more than 60min); SOX: Oxaliplatin: 130 mg/m2, administered intravenously, on the first day, once every three weeks, and every three weeks is a cycle; S-1: according to BSA (< <1.25 40 mg；; 1.25-1.5 50 mg； > >1.5 60 mg), oral administration, d1-d14 twice a day, 3 weeks as a cycle; Trazumab was administered intravenously, with an initial loading dose of 8 mg/kg and a subsequent dose of 6 mg/kg, with a cycle of 3 weeks
  Interventions: Drug: camrelizumab
- Cohort 2 (Active Comparator): camrelizumab was administered intravenously at a fixed dose of 200 mg, on the first day, once every 3 weeks, with a cycle of 3 weeks. Infusion for 30 min each time (no less than 20 min and no more than 60min); SOX: Oxaliplatin: 130 mg/m2, administered intravenously, on the first day, once every three weeks, and every three weeks is a cycle; S-1: according to BSA (< <1.25 40 mg；; 1.25-1.5 50 mg； > >1.5 60 mg), oral administration, d1-d14 twice a day, 3 weeks as a cycle;
  Interventions: Drug: camrelizumab

INTERVENTIONS:
Drug: camrelizumab — camrelizumab was administered intravenously at a fixed dose of 200 mg, on the first day, once every 3 weeks, with a cycle of 3 weeks. Infusion for 30 min each time (no less than 20 min and no more than 60min); SOX: Oxaliplatin: 130 mg/m2, administered intravenously, on the first day, once every three weeks, and every three weeks is a cycle; S-1: according to BSA (< <1.25 40 mg；; 1.25-1.5 50 mg； > >1.5 60 mg), oral administration, d1-d14 twice a day, 3 weeks as a cycle; Trastuzumab was administered intravenously, with an initial loading dose of 8 mg/kg and a subsequent dose of 6 mg/kg, with a cycle of 3 weeks.

SUMMARY:
A Study of the Advanced Adenocarcinoma of Stomach and Gastroesophageal Junction With Camrelizumab+SOX Control Camrelizumab+SOX+ Trastuzumab

DETAILED DESCRIPTION:
To observe the efficacy, safety, postoperative pathological remission rate and survival benefit of patients with HER-2 positive locally advanced adenocarcinoma of stomach and gastroesophageal junction treated with camrelizumab+SOX combined with trastuzumab or not.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-75 years old; Male or female; 2) Histopathological examination of gastroscopy biopsy confirmed adenocarcinoma of stomach and gastroesophageal junction; 3) Imaging (CT/MRI) and ultrasonic gastroscopy confirmed that: cT≥T2 and/or regional lymph node positive (N+); 4)HER-2 positive is the test result of IHC3+ or IHC2+/FISH+, and HER-2 test score standard refers to her-2 test guide for gastric cancer; 5)ECOG score: 0~1; 6) The expected survival time is ≥ 12 weeks; 7) The main organ functions meet the following criteria within 7 days before treatment:

  1. Blood routine examination standard (without blood transfusion within 14 days):

     Hb ≥ 90g/l; The absolute value of neutrophils (ANC) ≥ 1.5× 109/L; Platelet (PLT) ≥ 80× 109/L;
  2. Biochemical examination shall meet the following standards:

Total bilirubin (TBIL)≤1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× ULN; Serum creatinine (Cr)≤1.5 ULN or creatinine clearance rate (CCR) ≥ 60ml/min; (3) Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥ the lower limit of normal value (50%).

8) Women of childbearing age should agree to take contraceptive measures (such as intrauterine device, contraceptive pill or condom) during the study period and within 6 months after the end of the study; Serum or urine pregnancy test was negative within 7 days before the study was enrolled in the group, and it must be a non-lactating patient; Men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

9) Patients volunteered to participate in this study and signed an informed consent form;

Exclusion Criteria:

* 1) have had or are currently suffering from other malignant tumors within 5 years, except cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumor [Ta (non-invasive tumor), Tis (cancer in situ) and T1 (tumor infiltrating basement membrane)]; 2) Patients with distant metastasis and unable to undergo surgical resection; 3) Have a history of mental illness, or abuse of psychotropic drugs; 4) Subjects with diseases requiring systemic treatment with glucocorticoid (> 10 mg prednisone equivalent dose per day) or other immunosuppressive drugs within 14 days before the start of study treatment. In the absence of active autoimmune diseases, it is allowed to use inhaled or topical steroids > 10 mg daily prednisone equivalent dose and adrenal replacement steroid dose; 5) Those who have received any anti-tumor treatment in the past; 6) Participants who receive live/attenuated vaccines within 30 days; 7) Allergic reactions and adverse drug reactions:

  1. History of allergy to the ingredients of the study drug;
  2. Contraindications of any study drug (oxaliplatin or S-1) in chemotherapy regimen.

     8) Patients with any severe and/or uncontrollable diseases, including:

  <!-- -->

  1. Patients with hypertension who can't get good control after antihypertensive drug treatment (systolic blood pressure ≥180 mmHg, diastolic blood pressure ≥100 mmHg);
  2. Suffering from grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTc≥480 ms) and grade 2 or above congestive heart failure (new york Heart Association (NYHA) classification);
  3. Severe or uncontrolled disease or active infection (≥ CTCAE level 2 infection), which the researcher believes will increase the risks related to research participation, administration of research drugs or affect the ability of subjects to receive research drugs;
  4. Renal failure requires hemodialysis or peritoneal dialysis;
  5. those who have a history of immunodeficiency diseases, including HIV-positive or other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation; 9) Patients with a large number of ascites or poor ascites control; 10) preparing for or receiving allogeneic organ or allogeneic bone marrow transplantation, including liver transplantation; 11) Patients with brain metastasis; 12) Patients who are not suitable to participate according to the researcher's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate(pCR） | up to 2 years
  Refers to the absence of tumor cell residue in the primary tumor.

SECONDARY OUTCOMES:
Disease-free survival | up to 2 years
  Defined as postoperative disease-free subjects, starting from the time of postoperative baseline imaging evaluation to the time of disease recurrence or death.
Overall survival | up to 2 years
  defined as the time from the first medication to the death of a subject from any cause after enrollment. For the subjects who survived at the last contact, their total survival will be deleted on the last contact day.
Major pathological response rate | up to 2 years
  The survival tumor cells in the resected specimen were ≤10%.
R0 resection rate | up to 2 years
  There was no macroscopic tumor at the surgical margin, and the tumor cells at the surgical margin were negative within 1mm under microscope.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Tumor Hospital, Henan, China

IPD SHARING:
Plan to Share IPD: No